CLINICAL TRIAL: NCT01696019
Title: A Pilot Randomized Intervention Study of Physical Exercise and Social Engagement in Chinese Elders
Brief Title: Randomized Trial of Exercise and Social Interaction in a Community-Based Sample of Non-Demented Chinese Elders
Acronym: SCIBHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Byrd-ARG2007
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Cognitive Impairment; Dementia; Mild Cognitive Impairment; Alzheimer Disease
Keywords: magnetic resonance imaging; cognition; Tai Chi; physical exercise; mental exercise; intervention trial; prevention; dementia; Alzheimer disease; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease; Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fast walking (Experimental): Participants assigned to this group met with two group leaders three times per week in the morning in Jing An Park and were encouraged to walk quickly around a 400 meter circular route. Each session consisted of 10 minutes of warm-up stretching, 30 minutes of brisk walking, and 10 minutes of cool-down exercises. Prior to the first session, each participant was given a pedometer with their name on it. They were asked to take 100 steps and the sensitivity and positioning of the pedometer was adjusted to assure accurate measurement. At the termination of each session, the pedometers were collected and the number of steps taken by each participant at that session recorded. A record of the number of steps taken for every participant at each session over the 40 week period was maintained.
  Interventions: Other: Fast walking
- Tai Chi (Active Comparator): Participants assigned to this group met with a Tai Chi master and assistant three times per week in the morning in Jing An Park or at a nearby gymnasium depending on weather conditions. Each session included 20 min of warm-up exercises (lower back and hamstring stretching, gentle calisthenics, and balance training), 20 min of Tai Chi practice, and 10 min of cool-down exercises.
  Interventions: Other: Tai Chi
- Intellectual stimulation (Active Comparator): Participants assigned to this group met with a group leader and an assistant for one hour three times a week in the morning at the neighborhood community center. Although direction was initially given regarding subjects for discussion, the participants decided on their own to organize and select topics themselves.
  Interventions: Other: Intellectual stimulation
- Contact and testing only (Placebo Comparator): The fourth group received no intervention. Contact was maintained by phone during the intervention period to reduce dropout. Participants were called four times during the 40 weeks intervention period by the study coordinator.
  Interventions: Other: Contact and testing only

INTERVENTIONS:
Other: Fast walking — Participants assigned to this group met with two group leaders three times per week in the morning in Jing An Park and were encouraged to walk quickly around a 400 meter circular route. Each session consisted of 10 minutes of warm-up stretching, 30 minutes of brisk walking, and 10 minutes of cool-down exercises. Prior to the first session, each participant was given a pedometer with their name on it. They were asked to take 100 steps and the sensitivity and positioning of the pedometer was adjusted to assure accurate measurement. At the termination of each session, the pedometers were collected and the number of steps taken by each participant at that session recorded. A record of the number of steps taken for every participant at each session over the 40 week period was maintained.
  Arms: Fast walking
Other: Tai Chi — Participants assigned to this group met with a Tai Chi master and assistant three times per week in the morning in Jing An Park or at a nearby gymnasium depending on weather conditions. Each session included 20 min of warm-up exercises (lower back and hamstring stretching, gentle calisthenics, and balance training), 20 min of Tai Chi practice, and 10 min of cool-down exercises.
  Arms: Tai Chi
Other: Intellectual stimulation — Participants assigned to this group met with a group leader and an assistant for one hour three times a week in the morning at the neighborhood community center. Although direction was initially given regarding subjects for discussion, the participants decided on their own to organize and select topics themselves.
  Arms: Intellectual stimulation
Other: Contact and testing only
  Arms: Contact and testing only

SUMMARY:
A pilot randomized clinical trial was conducted in a random sample of 120 non-demented Chinese elders (ages 60-79) living in a defined community in Shanghai, China to compare the effects of interventions (fast walking, Tai Chi, group intellectual discussion) to no intervention with respect to change in cognition and whole brain volume determined by repeated neuropsychological batteries and MRI scans. Aims included determining the feasibility of recruiting and retaining a random sample of people age 60+ for such a trial as well as collection of preliminary data on the efficacy of the interventions. The long-term goal of this research program is to determine whether sustained physical and/or mental exercise interventions are efficacious in delaying the onset of dementia and to understand the role and mechanisms of brain growth in this process.

DETAILED DESCRIPTION:
Physical exercise has been shown to increase brain volume and improve cognition in randomized trials of non-demented elderly. Although greater social engagement was found to reduce dementia risk in observational studies, randomized trials of social interventions have not been reported. A representative sample of 120 elderly from Shanghai, China was randomized to four groups (Tai Chi, Walking, Social Interaction, No Intervention) for 40 weeks. Two MRI's were obtained, one before the intervention period, the other after. A neuropsychological battery was administered at baseline, 20 weeks and 40 weeks. Comparison of changes in brain volumes in intervention groups with the No Intervention group were assessed by t-tests. Time-intervention group interactions for neuropsychological measures were evaluated with repeated-measures mixed models.

ELIGIBILITY:
Inclusion Criteria:

* living in defined area
* either sex
* aged 60-79

Exclusion Criteria:

* history of stroke, Parkinson's disease or other neurologic disease
* inability to walk unassisted for two kilometers or maintain balance with feet side-by-side or semi-tandem for 10 seconds each
* education-adjusted Chinese Mini-Mental Examination score < 26 (to exclude individuals with dementia or moderate cognitive impairment
* cardiovascular or musculoskeletal conditions that would be contraindicated for the intervention programs
* contraindications for MRI
* diagnosis of any illness that would preclude participation in the full study
* regular vigorous exercise or Tai Chi practice.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance on battery of neuropsychological tests | Baseline, 4 months, 8 months
  A comprehensive battery of neuropsychological tests was administered by a psychometrist.

SECONDARY OUTCOMES:
Change in whole brain volume | Baseline, 8 months
  Structural MRIs were obtained at baseline and 8 months to provide data from which change in whole brain volume was determined.

CONTACTS AND LOCATIONS:
Overall Officials: James A Mortimer, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- Huashan Hospital, Shanghai, China

REFERENCES:
- [Result] Mortimer JA, Ding D, Borenstein AR, DeCarli C, Guo Q, Wu Y, Zhao Q, Chu S. Changes in brain volume and cognition in a randomized trial of exercise and social interaction in a community-based sample of non-demented Chinese elders. J Alzheimers Dis. 2012;30(4):757-66. doi: 10.3233/JAD-2012-120079. PMID 22451320